CLINICAL TRIAL: NCT02504580
Title: A Phase 2, Randomized, Pilot Study to Investigate the Safety, Efficacy, Pharmacokinetics and Bioavailability of HTX-011, HTX-002, or HTX-009 Administered Via Injection and/or Topical Application Following Unilateral Open Inguinal Herniorrhaphy
Brief Title: A Pilot Study to Investigate the Safety, Efficacy, Pharmacokinetics and Bioavailability of HTX-011, HTX-002, or HTX-009 Administered Via Injection and/or Topical Application Following Unilateral Open Inguinal Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-C2015-202
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (22):
- Part A, Cohort A (Experimental): HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg by injection.
  Interventions: Drug: HTX-011
- Part A, Cohort B (Experimental): HTX-011(bupivacaine/meloxicam), 400 mg/12 mg by injection.
  Interventions: Drug: HTX-011
- Part A, Cohort C (Experimental): HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg by instillation.
  Interventions: Drug: HTX-011
- Part A, Cohort D (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by instillation.
  Interventions: Drug: HTX-011
- Part A, Cohort E (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by injection and instillation (combination).
  Interventions: Drug: HTX-011
- Part A, Cohort F (Placebo Comparator): Saline placebo by injection.
  Interventions: Drug: Placebo
- Part B, Cohort A (Experimental): HTX-011A (bupivacaine/meloxicam), 200 mg/6 mg by injection.
  Interventions: Drug: HTX-011A
- Part B, Cohort B (Experimental): HTX-011A (bupivacaine/meloxicam) 400 mg12 mg by injection.
  Interventions: Drug: HTX-011A
- Part B, Cohort C (Experimental): HTX-011B (bupivacaine/meloxicam), 200 mg/6 mg by injection.
  Interventions: Drug: HTX-011B
- Part B, Cohort D (Experimental): HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg by injection.
  Interventions: Drug: HTX-011B
- Part B, Cohort E (Placebo Comparator): Saline placebo by injection.
  Interventions: Drug: Placebo
- Part C, Cohort A (Experimental): HTX-002, 200 mg by injection or instillation.
  Interventions: Drug: HTX-002
- Part B, Cohort F (Experimental): HTX-002, 400 mg by injection or instillation.
  Interventions: Drug: HTX-002
- Part C, Cohort B (Experimental): HTX-011B (bupivacaine/meloxicam), 200 mg/6 mg by instillation.
  Interventions: Drug: HTX-011B
- Part B, Cohort G (Experimental): HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg by instillation.
  Interventions: Drug: HTX-011B
- Part C, Cohort C (Placebo Comparator): Saline placebo by instillation.
  Interventions: Drug: Placebo
- Part C, Cohort D (Active Comparator): Bupivacaine HCI (Marcaine), 75 mg by injection.
  Interventions: Drug: Bupivacaine HCI (Marcaine)
- Part D, Cohort A (Experimental): HTX-011B (bupivacaine/meloxicam), 400 mg/13 mg via a combination of injection and instillation.
  Interventions: Drug: HTX-011B
- Part E, Cohort A (Experimental): HTX-009, 12 mg by injection and instillation (combination).
  Interventions: Drug: HTX-009
- Part F, Cohort A (Experimental): HTX-011B (bupivacaine/meloxicam), 300 mg/9 mg by instillation.
  Interventions: Drug: HTX-011B
- Part F, Cohort B (Experimental): Bupivacaine HCI (Marcaine), 75 mg by injection.
  Interventions: Drug: Bupivacaine HCI (Marcaine)
- Part F, Cohort C (Placebo Comparator): Saline placebo by injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam) by injection.
  Arms: Part A, Cohort A; Part A, Cohort B; Part A, Cohort C; Part A, Cohort D; Part A, Cohort E
Drug: Placebo — Saline placebo by injection.
  Arms: Part A, Cohort F; Part B, Cohort E; Part C, Cohort C; Part F, Cohort C
Drug: HTX-002 — HTX-002, by injection or instillation (pooled).
  Arms: Part B, Cohort F; Part C, Cohort A
Drug: Bupivacaine HCI (Marcaine) — Bupivacaine HCI (Marcaine) by injection.
  Arms: Part C, Cohort D; Part F, Cohort B
Drug: HTX-011A — HTX-011A (bupivacaine/meloxicam) by injection.
  Arms: Part B, Cohort A; Part B, Cohort B
Drug: HTX-011B — HTX-011B (bupivacaine/meloxicam) by injection, instillation or combination.
  Arms: Part B, Cohort C; Part B, Cohort D; Part B, Cohort G; Part C, Cohort B; Part D, Cohort A; Part F, Cohort A
Drug: HTX-009 — HTX-009 by injection and instillation (combination).
  Arms: Part E, Cohort A

SUMMARY:
A Phase 2, Randomized, Pilot Study to Investigate the Safety, Efficacy, Pharmacokinetics and Bioavailability of HTX-011, HTX-002, or HTX-009 Administered Via Injection and/or Topical Application Following Unilateral Open Inguinal Herniorrhaphy

DETAILED DESCRIPTION:
This study includes multiple formulations for formulation selection of the fixed-combination product and for the factorial design assessment of the contribution of each component. HTX-011 is the initial formulation studied (HTX-011-19). HTX-011A is the second formulation studied (HTX-011-49). HTX-011B is the final formulation studied (HTX-011-56), which was also included in subsequent Phase 2b and Phase 3 studies. For the factorial design assessment, HTX-002, a bupivacaine-only formulation in the same HTX-011 proprietary polymer, and HTX-009, a meloxicam-only formulation in the same HTX-011 proprietary polymer, were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female 18 years of age or older.
2. Female subjects are eligible only if all of the following apply:

   Not pregnant (female subject of child bearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test before surgery)
   * Not lactating
   * Not planning to become pregnant during the study
   * Be surgically sterile; or at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study and for 30 days from completion of the study

   Male:

   o Must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 1 week after the administration of study medication.
3. Plan to undergo a unilateral inguinal herniorrhaphy
4. Have the ability and be willing to comply with the study procedures
5. Must be able to understand study procedures and give informed consent for the conduct for all study procedures, using an IRB approved consent form.

Exclusion Criteria:

1. Unwilling to sign informed consent or not willing or able to complete all study procedures
2. Have a contraindication or be allergic to any medication to be used during the trial period
3. Have clinically significant cardiac abnormalities, that in the opinion of the investigator would pose a health risk to the subject should they participate in the trial
4. Have American Society of Anesthesiologists (ASA) Physical Status classification system category 4 or greater (Appendix E)
5. Have clinically significant renal or hepatic abnormalities (defined as an AST or ALT > 3x ULN, creatinine > 2x ULN)
6. Have another painful condition that may confound pain assessments
7. Have another surgery planned within 30 days of procedure, or presents with bilateral or recurrent inguinal hernia, other hernia presentations, or hernias with large scrotal component that would be difficult to reduce surgically
8. Have a known or suspected history of alcohol or drug abuse, or a positive drug screen
9. Currently taking analgesics for a chronically painful condition, or has taken long acting opioids within 3 days of surgery, or taken any opioids within 24 hours of surgery
10. Subjects with documented sleep apnea or are on home continuous positive airway pressure (CPAP)
11. Female subjects who are pregnant (positive pregnancy test at screening or on the day of surgery)
12. Subjects who are receiving oxygen therapy at the time of screening
13. Have participated in a clinical trial within 30 days of planned surgery
14. Have a body mass index (BMI) > 39 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anaheim, California
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study HTX-011-202 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- Part A, Cohort A: HTX-011: HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg by injection.
- Part A, Cohort B: HTX-011: HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by injection.
- Part A, Cohort C: HTX-011: HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg by instillation.
- Part A, Cohort D: HTX-011: HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by instillation.
- Part A, Cohort E: HTX-011: HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by injection and instillation (combination).
- Part A, Cohort F: Saline Placebo; Parts B/C/D/E/F/G: Saline Placebo: Saline placebo by injection.
- Parts B/C/D/E/F/G: HTX-011A: HTX-011A (bupivacaine/meloxicam), 200-400 mg/6-12 mg by injection.
- Parts B/C/D/E/F/G: HTX-011B: HTX-011B (bupivacaine/meloxicam) 200-400 mg/6-12 mg by injection, instillation or combination (pooled).
- Parts B/C/D/E/F/G: HTX-011-002: HTX-002, 200-400 mg by injection or instillation (pooled).
- Parts B/C/D/E/F/G: HTX-009: HTX-009, 12 mg by injection and instillation (combination).
- Parts B/C/D/E/F/G: Bupivacaine (Marcaine): Bupivacaine HCI, 75 mg by injection.
Period: Overall Study
Arm/Group | Part A, Cohort A: HTX-011 | Part A, Cohort B: HTX-011 | Part A, Cohort C: HTX-011 | Part A, Cohort D: HTX-011 | Part A, Cohort E: HTX-011 | Part A, Cohort F: Saline Placebo | Parts B/C/D/E/F/G: HTX-011A | Parts B/C/D/E/F/G: HTX-011B | Parts B/C/D/E/F/G: HTX-011-002 | Parts B/C/D/E/F/G: HTX-009 | Parts B/C/D/E/F/G: Bupivacaine (Marcaine) | Parts B/C/D/E/F/G: Saline Placebo
Started | 19 | 17 | 16 | 20 | 17 | 18 | 40 | 131 | 52 | 18 | 32 | 83
Completed | 18 | 16 | 16 | 18 | 16 | 17 | 39 | 129 | 52 | 18 | 32 | 81
Not Completed | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 2
Not completed — Other | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 2
Not completed — Subject refusal to continue | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study HTX-011-202 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- Part A, Cohorts A, B C, D, E: HTX-011: HTX-011 (bupivacaine/meloxicam), 200-400 mg/6-12 mg by injection, instillation or combination (pooled).
- Part B/C/D/E/F/G: HTX-011A: HTX-011A (bupivacaine/meloxicam), 200-400 mg/6-12 mg by injection.
- Parts B/C/D/E/F/G: HTX-002: HTX-002, 200-400 mg by injection or instillation (pooled).
- Parts B/C/D/E/F/G: HTX-011B: HTX-011B (bupivacaine/meloxicam), 200-400 mg/6-12 mg by injection, instillation or combination (pooled).
- Parts B/C/D/E/F/G: Bupivacaine (Marcaine: Bupivacaine HCI, 75 mg by injection.
- Parts A/B/C/D/E/F/G: Saline Placebo: Saline placebo by injection.
- Total: Total of all reporting groups
Arm/Group | Part A, Cohorts A, B C, D, E: HTX-011 | Part A, Cohort F: Saline Placebo | Part B/C/D/E/F/G: HTX-011A | Parts B/C/D/E/F/G: HTX-002 | Parts B/C/D/E/F/G: HTX-011B | Parts B/C/D/E/F/G: HTX-009 | Parts B/C/D/E/F/G: Bupivacaine (Marcaine | Parts A/B/C/D/E/F/G: Saline Placebo | Total
Number analyzed (Participants) | 89 | 18 | 39 | 51 | 131 | 18 | 32 | 85 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (12.56) | 46.5 (13.99) | 50.8 (9.99) | 46.8 (14.26) | 45.6 (13.30) | 49.8 (10.73) | 41.7 (12.74) | 46.0 (12.40) | 46.1 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 12
  Male | 84 | 18 | 39 | 49 | 129 | 17 | 31 | 84 | 451
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 7 | 13 | 21 | 57 | 4 | 11 | 36 | 191
  Not Hispanic or Latino | 47 | 11 | 26 | 30 | 74 | 14 | 21 | 49 | 272
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 0 | 6 | 6 | 11 | 4 | 4 | 14 | 57
  White | 77 | 18 | 33 | 45 | 112 | 13 | 27 | 70 | 395
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 89 | 18 | 39 | 51 | 131 | 18 | 32 | 85 | 463

OUTCOME MEASURES:

1. Primary Outcome: Mean Summed Pain Intensity (SPI) Score.
Description: The SPI is derived by summing the pain intensity score weighted by the scheduled time duration. SPI0-24 will be calculated by summing the Pain intensity (PI) score at the relevant time points weighted by the scheduled time duration since the prior PI assessment as follows: SPI0-24= PI1+PI2+2*PI4+2*PI6+2*PI8+2*PI10+2*PI12+2*PI14+4*PI18+6*PI24. Min = 0 (if PI=0 at every time) and Max = 240 (if PI=10 at every time).
Time Frame: 24 hours
Population: mITT Population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- HTX-011: 200 mg: HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg by injection or instillation.
- HTX-011: 400 mg: HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg by injection or instillation or combination.
- HTX-011A: 200 mg: HTX-011A (bupivacaine/meloxicam), 200 mg/6 mg by injection.
- HTX-011A: 400 mg: HTX-011A (bupivacaine/meloxicam), 400 mg/12 mg by injection.
- HTX-011B: 200 mg: HTX-011B (bupivacaine/meloxicam), 200 mg/6 mg by injection or instillation (pooled).
- HTX-011B: 300 mg: HTX-011B (bupivacaine/meloxicam), 300 mg/9 mg by instillation.
- HTX-011B: 400 mg: HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg by injection, instillation or combination (pooled).
- HTX-002: 200 mg: HTX-002, 200 by injection or instillation.
- HTX-002: 400 mg: HTX-002, 400 mg by injection or instillation
- HTX-009: 12 mg: HTX-009, 12 mg by injection and instillation (combination).
- Saline Placebo: Saline placebo by injection or combination.
- Bupivacaine HCI: Bupivacaine HCI, 75 mg by injection.
Arm/Group | HTX-011: 200 mg | HTX-011: 400 mg | HTX-011A: 200 mg | HTX-011A: 400 mg | HTX-011B: 200 mg | HTX-011B: 300 mg | HTX-011B: 400 mg | HTX-002: 200 mg | HTX-002: 400 mg | HTX-009: 12 mg | Saline Placebo | Bupivacaine HCI
Number analyzed (Participants) | 35 | 54 | 21 | 18 | 31 | 16 | 84 | 22 | 30 | 18 | 83 | 32
Units on a scale | 83.71 (45.996) | 77.63 (40.679) | 95.24 (50.135) | 89.28 (59.403) | 97.16 (49.093) | 73.81 (50.572) | 86.61 (40.091) | 99.82 (41.433) | 99.53 (45.415) | 118.22 (26.399) | 121.93 (48.239) | 108.72 (37.552)

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: Study HTX-011-202 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- Part A: Saline Placebo; Parts B/C/D/E/F/G: Saline Placebo: Saline placebo by injection.
- Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-011A: HTX-011A (bupivacaine/meloxicam), 200-400 mg/6-12 mg by injection.
- Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-002: HTX-002, 200-400 mg by injection or instillation (pooled).
- Parts B/C/D/E/F/G: HTX-011-009: HTX-009, 12 mg by injection and instillation (combination).
- Parts B/C/D/E/F/G: Bupivacaine HCI (Marcaine): Bupivacaine HCI, 75 mg by injection.
Arm/Group | Part A, Cohorts A, B C, D, E: HTX-011 | Part A: Saline Placebo | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-011A | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-002 | Parts B/C/D/E/F/G: HTX-011B | Parts B/C/D/E/F/G: HTX-011-009 | Parts B/C/D/E/F/G: Bupivacaine HCI (Marcaine) | Parts B/C/D/E/F/G: Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/18 | 0/39 | 0/51 | 0/131 | 0/18 | 0/32 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/18 | 0/39 | 0/51 | 2/131 | 2/18 | 1/32 | 1/85
Other Adverse Events (participants affected / at risk) | 56/89 | 13/18 | 20/39 | 28/51 | 85/131 | 13/18 | 19/32 | 52/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohorts A, B C, D, E: HTX-011 (N=89) | Part A: Saline Placebo (N=18) | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-011A (N=39) | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-002 (N=51) | Parts B/C/D/E/F/G: HTX-011B (N=131) | Parts B/C/D/E/F/G: HTX-011-009 (N=18) | Parts B/C/D/E/F/G: Bupivacaine HCI (Marcaine) (N=32) | Parts B/C/D/E/F/G: Saline Placebo (N=85)
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohorts A, B C, D, E: HTX-011 (N=89) | Part A: Saline Placebo (N=18) | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-011A (N=39) | Part B/C/D/E/F/G: Part B/C/D/E/F/G: HTX-002 (N=51) | Parts B/C/D/E/F/G: HTX-011B (N=131) | Parts B/C/D/E/F/G: HTX-011-009 (N=18) | Parts B/C/D/E/F/G: Bupivacaine HCI (Marcaine) (N=32) | Parts B/C/D/E/F/G: Saline Placebo (N=85)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 0 | 3 | 6 | 24 | 4 | 4 | 7
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 1 | 7 | 1 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 10 | 1 | 2 | 1 | 7 | 2 | 2 | 6
Tachycardia (Cardiac disorders) | 4 | 4 | 4 | 0 | 7 | 2 | 2 | 5
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 7 | 3 | 1 | 0 | 2 | 0 | 1 | 5
Hypotension (Vascular disorders) | 3 | 0 | 0 | 1 | 9 | 0 | 1 | 4
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 28 | 6 | 9 | 14 | 41 | 8 | 8 | 28
Nausea (Gastrointestinal disorders) | 8 | 6 | 2 | 10 | 30 | 4 | 6 | 19
Vomiting (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 7 | 2 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 9 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1 | 4 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 2 | 7 | 0 | 2 | 1
Scrotal mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Induration (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spermatic cord disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT02504580/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02504580/SAP_001.pdf